CLINICAL TRIAL: NCT05705102
Title: Time for a DIagnostic Paradigm Shift From ST-elevation/Non-ST-elevation to OCClUsion/Non-occLusion Myocardial infarcTion?
Brief Title: Time for a Paradigm Shift: STEMI/NSTEMI to OMI/NOMI ?
Acronym: DIFOCCULT-2
Status: Terminated | Type: Observational
Why Stopped: Problems due to retrospective data acquisition
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Emre Aslanger, Associate Professor, Marmara University
Other Study IDs: MarmaraCard002
Record Dates: First submitted 2023-01-21; First posted 2023-01-30 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Myocardial Infarction; Myocardial Ischemia
Keywords: acute coronary occlusion; electrocardiography; myocardial infarction; ST-segment elevation
MeSH Terms: conditions — Myocardial Infarction; Myocardial Ischemia | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OMI/NOMI group: In this group, the patients will be managed according to OMI/NOMI paradigm. OMI patients, even without STEMI criteria, will be taken immediately to the cath lab.
  Interventions: Other: Coronary intervention
- STEMI/NSTEMI group: Standard care
  Interventions: Other: Coronary intervention

INTERVENTIONS:
Other: Coronary intervention — Coronary intervention will be done immediately in patients with OMI (even STEMI criteria are negative), instead of waiting for <24h.

SUMMARY:
The current ST-segment elevation (STEMI)/non-STEMI treatment paradigm misses nearly one fourth of acute coronary occlusions (ACO) that needs immediately reperfusion. Many of these cases can be recognized by subtle changes on ECG, but the current STEMI criteria do not include them. The investigators of this research believe a new occlusive/non-occlusive myocardial infarction (OMI/NOMI) approach will be superior to the established STEMI/non-STEMI paradigm in early detection of ACO, limiting infarct size, reducing re-hospitalizations and most important of all, reducing mortality.

DETAILED DESCRIPTION:
The patients with acute coronary occlusion (ACO) or potentially imminent occlusion, with insufficient collateral circulation, have myocardium that is at risk of infarction unless they undergo immediate reperfusion via thrombolytics or percutaneous coronary intervention (PCI). One of the most important tasks in emergency cardiology is to immediately identify acute coronary occlusion (ACO) myocardial infarction (OMI) among all patients who present with symptoms compatible with acute myocardial infarction (MI), and distinguish them from those without MI, and from those with MI that does not have ongoing myocyte loss (Non-OMI, or NOMI) who can be managed with medical therapy and for whom potentially harmful invasive interventions can be deferred. The electrocardiogram (ECG) plays a central role in this process.

The presence or absence of ST-segment elevation (STE) is principally used to define patients who need emergent coronary revascularization, since subgroup analyses of the Fibrinolytic Therapy Trialists' (FTT) meta-analysis indicated that patients with STE on ECG gain a slightly better survival benefit from emergent reperfusion. After fine-tuning of STE cutoffs used in this analysis, universally agreed STEMI criteria became the current guideline-supported ECG paradigm.

However, the evidence accumulated in the past 20 years indicate that there is still room for substantial improvement. Although patients with ACO are the group that is believed to benefit from emergent reperfusion therapy, fibrinolytic studies did not investigate the presence or absence of ACO among enrolled patients. Moreover, they did not specifically focus on ECG findings, including STE; four of the nine trials even did not use ECG for enrollment, and the remaining five defined their version of STE with varying cutoffs, and without specified measurement methods. To reconcile different STE criteria used in various studies, several investigators compared STE in normal subjects and patients with MI. However, none of the studies cited in the current universal definition of MI used ACO on angiography as an endpoint, so these criteria were actually not designed to differentiate STEMI from non-STEMI.

In the past 20 years, several investigators, including this group, have demonstrated that factors other than STE, including STE of magnitude less than those recommended by the guidelines (but in combination with other features), can help in diagnosing ACO or excluding it. Proportionality, which is unfortunately completely absent in the STEMI criteria, is a common factor in most of these studies: proportionality is the idea that any amount of STE or ST-segment depression (STD), or T-wave size, must be assessed relative to the QRS amplitude. Many other clues should also be taken into account when differentiating STE due to ACO from other causes of STE, which has been described in detail in recent reviews published by our group.

Studies show current STEMI criteria miss nearly one-third of ACO with the result that this unfortunate group of patients, labeled as non-STEMI, are deprived of emergent reperfusion therapy. Many studies showed that approximately one third to one-fifth of the patients with ACO had equal to or less than 1 mm of STE, hyperacute T-waves, non-contiguous STE patterns, etc. These patients are unfortunately deprived of emergent reperfusion therapy and ACO is only found after rising troponin level identifies them as having MI and they undergo a next-day angiogram. Furthermore, this proportion may be underestimated, since a large percentage of total thrombotic occlusions spontaneously reperfuse by this time; unfortunately, only after a substantial loss of myocardium. These findings are highly relevant and important, as those with unrecognized ACO had higher short and long-term risk of mortality.

Recently, the DIagnostic accuracy oF electrocardiogram for acute coronary OCClUsion resuLTing in myocardial infarction (DIFOCCULT) study [1], compared OMI/non-OMI approach with STEMI/non-STEMI paradigm. This is the largest study specifically designed to question the STEMI/non-STEMI paradigm, in which a set of predefined ECG findings in addition to STEMI criteria were used, and the final outcome was a composite ACO endpoint. In accordance with the previous observations, over one-fourth of the patients initially classified as having non-STEMI were re-classified by the ECG reviewers, blinded to all outcome data, as having OMI. This subgroup had a higher frequency of ACO, myocardial damage, and both in-hospital and long-term mortality compared to the non-OMI group. The OMI/non-OMI approach to the ECG had a superior diagnostic accuracy compared to the STE/non-STEMI approach in the prediction of both ACO and long-term mortality.

Similarly, another retrospective case-control study [2] of 808 patients with suspected acute coronary syndrome (ACS) symptoms compared the accuracy of STEMI criteria vs. structured expert ECG interpretation which incorporates other findings of OMI including hyper-acute T-waves, STD of posterior OMI, STE less than the STEMI criteria cutoffs, etc. STEMI (-) OMI patients had similar infarct size measured by peak troponin but greater delays to angiography compared with the STEMI (+) OMI patients. Of the 808 patients, 49% had MI (33% OMI; 16% NOMI). Sensitivity, specificity, and accuracy of STEMI criteria vs Expert 1 for OMI among all 808 patients were 41% vs 86%, 94% vs 91%, and 77% vs 89%, and for Expert 2 among 250 patients were 36% vs 80%, 91% vs 92%, and 76% vs 89%. OMIs were correctly diagnosed a median of 1.5 hours (mean 3.0 hours) earlier by structured expert ECG interpretation than by STEMI criteria, or by angiogram if the ECG never met STEMI criteria.

Lastly, the STEMI/NSTEMI vs. OMI/NOMI paradigm were compared in 467 consecutive high/risk acute coronary syndrome patients [3]. Among the 108 patients with OMI, only 60% had any ECG meeting STEMI criteria. STEMI (-) OMI patients had similar peak troponins, wall motion abnormalities, left ventricular ejection fraction (LVEF) and clinical outcomes as compared with the STEMI (+) OMI patients, but were much less likely to receive emergent catheterization.

These data support the notion that the STEMI (-) but OMI (+) patients likely represent a missed opportunity under the STEMI/NSTEMI paradigm. A new OMI/NOMI approach has the potential of being the next significant improvement in modern MI care.

The hypothesis of this study is that the new OMI/NOMI approach will be superior to the established STEMI/NSTEMI paradigm in early detection of ACO, limiting infarct size, reducing rehospitalizations and most important of all, reducing mortality.

The adult patients (age >18 years) who are admitted to the emergency department with a clinical picture compatible with acute coronary syndrome will be screened for enrollment into the study. If any ECG in the emergency department is recognized as OMI/STEMI (according to the treating provider) or if the troponins are elevated, the patient will be enrolled into the study.

Before the study a detailed briefing will be done to the interventional cardiologists who will form the intervention groups.

Although the STEMI/NSTEMI approach is the current norm (a diagnosis of STEMI requires emergent catheterization, whereas the patients with NSTEMI are stabilized first and then electively undergo catheterization unless there are high-risk features), it would be unethical for a ECG reviewer, who is trained in recognizing the signs of ACO not fulfilling the current STEMI criteria, to suspend emergent reperfusion therapy after an OMI diagnosis has been made. Therefore, the ECG interpreters who are trained in OMI diagnosis cannot be randomized to STEMI/NSTEMI versus OMI/NOMI approaches. Hence, the groups will be randomized in the following fashion: A OMI/NOMI and a STEMI/NSTEMI intervention group will be formed. Intervention group 1 will be encouraged to use OMI/NOMI approach in patients with suspected acute coronary syndrome, and group 2 will use the current STEMI/NSTEMI approach.

The ECG interpreters (who contact the patient first and decide the treatment style, according to the center this can be either an emergency physician or a cardiologist) in both groups will be ensured to have a similar experience in terms of years of training. The ECG interpreter will thus elect to go for catheterization based on his/her ECG approach and, whether that is by OMI or STEMI paradigm, the patient will be enrolled accordingly and the reason for proceeding to the catheterization laboratory will be written on the study form. The interventional cardiologists in both groups will be ensured to have a similar experience level (in terms of years of training, and angiography and primary PCI counts in the past year). In the STEMI/NSTEMI arm, the contributors will blindly continue their practice, the ECG interpretation and decision to activate the catheterization laboratory will be done as usual. In the OMI/NOMI arm, an intensive course on ECG diagnosis of OMI using previously published algorithms and ECGs will be provided [4, 5]. After these two groups are formed, the patients will be block-randomized into STEMI/NSTEMI and OMI/NOMI cohorts according to the team on-duty. No intervention to the decisions will be done during the study process.

The STEMI/NSTEMI group will use the following criteria for the diagnosis of STEMI: (1) New ST-segment elevation at the J-point in two contiguous leads with the cut-point: ≥ 1 mm in all leads other than leads V2-V3 where the following cut-points apply: ≥2 mm in men ≥40 years; ≥2.5 mm in men <40 years, or ≥1.5 mm in women regardless of age, and (2) a peak troponin level above 99th percentile and (3) a clinical picture compatible with acute coronary syndrome. If the decision to proceed to the cath lab was done only with the first criterion, the participant will remain in the study, even if the second criterion is not met. The patients meeting only criteria (2) and (3) will be classified as NSTEMI.

In the OMI/NOMI group, the algorithm defined in the DIFOCCULT trial [1, 4, 5] will be used for ECG diagnosis (1). Additionally (2) a peak troponin level above 99th percentile and (3) a clinical picture compatible with acute coronary syndrome will be required. If the decision to proceed emergently to the cath lab was done only with the first criterion, the participant will remain in the study, even if the second criterion is not met. The patients who do not meet ECG-OMI criteria will be classified as NOMI, if: (1) a peak troponin level above 99th percentile and (2) a clinical picture compatible with acute coronary syndrome is present.

STEMI and OMI patients (will be taken as STEMI equivalents) will be managed according to the current STEMI guidelines, whereas NSTEMI and NOMI patients are managed according to the current NSTEMI guidelines. A separate diagnostic group with 'probable OMI' and 'high-risk STEMI' is also allowed for patients who do not fulfil STEMI/OMI criteria but need urgent catheterization for other high-risk features or high clinical suspicion for having an ACO. These patients will also be managed according to the current guidelines. However, patients will be excluded from analysis if their early catheterization is based solely on social or logistical considerations, and not based on the medical need. For example, a patient would be excluded if he/she is brought to the cath lab early based on the immediate availability of cath lab or because the patient is already scheduled for elective coronary angiography.

No other intervention will be done during study. After the patient enrollment period, data will be retrieved from the system and will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Clinical picture compatible with acute coronary syndrome AND recognized as OMI/STEMI (according to the treating provider) or cardiac high-sensitive troponins levels are elevated

Exclusion Criteria:

* Unable to acquire ECG

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The adult patients who are admitted to the emergency department with a clinical picture compatible with acute coronary syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Mortality | One year
  Mortality
Mortality in OMI (+) but STEMI (-) patients | One year
  Mortality in OMI (+) but STEMI (-) patients

SECONDARY OUTCOMES:
ACO | At index hospitalization (<7 day)
  Acute coronary occlusion on angiogram
Infarct size | At index hospitalization (<7 day)
  Infarct size by 72-hour peak troponin level
Left ventricular function | At index hospitalization (<7 day)
  Left ventricular function by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Emre Aslanger, Principal Investigator — Marmara University
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aslanger EK, Yildirimturk O, Simsek B, Bozbeyoglu E, Simsek MA, Yucel Karabay C, Smith SW, Degertekin M. DIagnostic accuracy oF electrocardiogram for acute coronary OCClUsion resuLTing in myocardial infarction (DIFOCCULT Study). Int J Cardiol Heart Vasc. 2020 Jul 30;30:100603. doi: 10.1016/j.ijcha.2020.100603. eCollection 2020 Oct. PMID 32775606
- [Background] Pendell Meyers H, Bracey A, Lee D, Lichtenheld A, Li WJ, Singer DD, Rollins Z, Kane JA, Dodd KW, Meyers KE, Shroff GR, Singer AJ, Smith SW. Accuracy of OMI ECG findings versus STEMI criteria for diagnosis of acute coronary occlusion myocardial infarction. Int J Cardiol Heart Vasc. 2021 Apr 12;33:100767. doi: 10.1016/j.ijcha.2021.100767. eCollection 2021 Apr. PMID 33912650
- [Background] Meyers HP, Bracey A, Lee D, Lichtenheld A, Li WJ, Singer DD, Kane JA, Dodd KW, Meyers KE, Thode HC, Shroff GR, Singer AJ, Smith SW. Comparison of the ST-Elevation Myocardial Infarction (STEMI) vs. NSTEMI and Occlusion MI (OMI) vs. NOMI Paradigms of Acute MI. J Emerg Med. 2021 Mar;60(3):273-284. doi: 10.1016/j.jemermed.2020.10.026. Epub 2020 Dec 9. PMID 33308915
- [Background] Aslanger EK, Meyers PH, Smith SW. STEMI: A transitional fossil in MI classification? J Electrocardiol. 2021 Mar-Apr;65:163-169. doi: 10.1016/j.jelectrocard.2021.02.001. Epub 2021 Feb 13. PMID 33640636
- [Background] Aslanger EK, Meyers HP, Smith SW. Recognizing electrocardiographically subtle occlusion myocardial infarction and differentiating it from mimics: Ten steps to or away from cath lab. Turk Kardiyol Dern Ars. 2021 Sep;49(6):488-500. doi: 10.5543/tkda.2021.21026. PMID 34523597